CLINICAL TRIAL: NCT00363701
Title: With-Drawal Study of Proton-Pump-Inhibitors in Patients From Primary Care Who Have Previously Been Treated on a Long-Term Basis
Brief Title: Study of Long-Term Use of Proton-Pump-Inhibitors in General Practice
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Last update posted 2006-08-15 (Estimated); Status verified 2006-08

CONDITIONS: Dyspepsia; Gastroesophageal Refluxdisease; Ulcer
Keywords: Protonpumpinhibitors; withdrawal; longterm treatment; dyspepsia; functional dyspepsia; gastrooesophageal reflux; upper endoscopy
MeSH Terms: conditions — Dyspepsia; Ulcer; Gastroesophageal Reflux | interventions — Esomeprazole

INTERVENTIONS:
Drug: esomeprazole

SUMMARY:
The primary purpose of the study is to determine the effect of esomeprazole compared to placebo in patients from general practice who have previously been treated with proton-pump-inhibitors (PPI) and who have no upper endoscopic findings.

DETAILED DESCRIPTION:
The majority of patients with dyspepsia are treated in primary care with acid-suppressive therapy for shorter or longer periods of time on the assumption that the patients´ symptoms are related to the production of acid in the stomach.

In about half of the dyspeptic patients there is no structural or biochemical explanation for their symptoms. These patients suffer from functional dyspepsia.

Treatment with proton-pump-inhibitors is effective in treating patients with gastroesophageal refluxdisease or ulcers. It is however controversial if acid-suppressive treatment is effective in the large group of patients with functional dyspepsia. Previous studies have shown no or very modest effect with a very high placeboresponse rate of 40-50%.

In primary care patients with upper abdominal symptoms are often treated with PPI as a diagnostic tool. If the treatment is effective continued or repeated treatment with PPI is often favored. However some of the patients must experience the abovementioned placebo-effect. These patients may end up being treated with PPI long-term on uncertain indication.

We wish to investigate the consequences of withdrawing treatment with PPI in patients from general practice who have previously been treated long-term.

An upper endoscopy is performed in patients who experience upper abdominal symptoms after withdrawal of treatment.If the endoscopy is normal patients are randomised to 1 week treatment with either esomeprazole or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with PPI in at least 4 months out of the preceding 12.
* Use of PPI in the preceding 10 out of 30 days before inclusion
* Age above 18 years

Exclusion Criteria:

* Erosive Esophagitis
* PPI-treatment as prophylaxis against gastrointestinal bleeding
* PPI-treatment as prophylaxis against ulcers
* PPI-treatment as prophylaxis because of NSAID-treatment
* Pregnant or lactating women
* Previous upper GI surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2006-08; Study Completion 2008-02

PRIMARY OUTCOMES:
Comparison of the effect of treatment in one week with esomeprazole and placebo measured as symptomscore in patientdiary.

SECONDARY OUTCOMES:
Fraction of patients who are willing to withdraw treatment with PPI
Fraction of patients who experience symptoms after withdrawal of treatment.
Description of endoscopic findings in patients who have previously been treated with PPI long-term and who after withdrawal are symptomatic
Length of time from withdrawal till symptoms arise
Correlation between levels of gastrin and CgA and time till symptoms arise
Investigators and patients ability to distinguish between active and placebo treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bytzer, ass. professor, ph.d, Principal Investigator — Glostrup University Hospital
Locations (1):
- Department of gastroenterology, Glostrup University Hospital, Glostrup Municipality, Denmark